CLINICAL TRIAL: NCT02722174
Title: Fingerprinting of Impulsivity in Four Diagnostic and Statistical Manual of Mental Disorders, Version 5 (DSM-5) Psychiatric Disorders That Have Been Clinically Associated With Impulsivity Using a Battery of Questionnaires and Behavioral Laboratory Tests
Brief Title: Fingerprinting of Impulsivity
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 352.2073
Record Dates: First submitted 2016-03-23; First posted 2016-03-29 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Impulse Control Disorders
MeSH Terms: conditions — Disruptive, Impulse Control, and Conduct Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (6):
- BED: Binge Eating Disorder
- ADHD: Attention Deficit Hyperactivity Disorder
- SUD, cocaine subtype: Stimulant Use Disorder, cocaine subtype
- BPD: Borderline Personality Disorder
- BPD, Cohort 2: Borderline Personality Disorder, Cohort 2
- HC: Healthy Controls

SUMMARY:
The study aims to examine a battery of behavioral and questionnaire measures in 4 disorders clinically associated with impulsivity and in health controls, to: 1) investigate if the different populations have a distinct behavioral profile, and 2) to investigate if there are specific measures that are reliable and sensitive measures of impulsivity across diagnoses.

ELIGIBILITY:
Inclusion criteria:

All cohorts:

- Males and females ages 18-50.

Healthy Control cohort:

- Volunteers in generally good Psychiatric and non-Psychiatric medical health

Borderline Personality Disorder (2 cohorts):

- Subjects who meet Diagnostic and Statistical Manual of Mental Disorders-V (DSM-V) criteria for Borderline Personality Disorder

Binge Eating Disorder cohort:

- Subjects who meet DSM-V criteria for Binge Eating Disorder.

Stimulant Use Disorder cohort:

- Subjects who meet DSM-V criteria for current Stimulant Use Disorder, subtype cocaine, moderate or severe use

Attention Deficit Hyperactivity Disorder cohort:

- Subjects who meet DSM-V criteria for adult Attention Deficit Hyperactivity Disorder

Exclusion criteria:

General:

* Positive breathalyzer test for alcohol at any study visit
* History of clinically significant neurologic disorders or head trauma with loss of consciousness greater than 30 minutes
* Clinically significant non-psychiatric medical disorder requiring ongoing treatment as judged by the investigator.
* Unwillingness or inability to sign a written informed consent form
* Pregnancy as assessed by a urine test for ß-Human Chorionic Gonadotropin (ß-HCG) at screening visit
* Medical or physical contraindications for participation (see below), based on medical history interview, as judged by the investigator
* Unwilling to refrain from tobacco use one hour prior to testing until after conclusion of testing

Healthy Controls:

* Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 diagnoses of Personality Disorders (based on Structured Clinical Interview for DSM-IV (SCID)-II)
* DSM-5 diagnoses based on the SCID-I (including the eating disorders and Attention Deficit Hyperactivity Disorder (ADHD) module)
* History of arrest or incarceration
* Positive urine drug screen for cannabis, cocaine, opioids, amphetamine, and benzodiazepines at any visit
* Current Tobacco Users

Borderline Personality Disorder Subjects:

* DSM-5 diagnoses other than: Tobacco Use Disorder, Major Depressive Disorder (Mild Subtype), Generalized Anxiety Disorder (in remission), Post-Traumatic Stress Disorder (in remission), Major Depressive Disorder (Moderate or Severe Subtype, in remission), or Substance use disorder (Mild subtype, in remission)
* DSM-5 Personality Disorder other than Cluster B Personality disorders.
* Positive urine drug screen for cocaine, opioids, amphetamine, and benzodiazepines at any visit
* Antipsychotic medication or mood stabilizers taken within the last 30 days or change in antidepressant medication within the last 30 days.

Binge Eating Disorder Subjects:

* DSM-5 diagnoses other than: Binge Eating Disorder (current bulimia also excluded), Tobacco Use Disorder, Major Depressive Disorder (in remission), Generalized Anxiety Disorder (in remission), Post-Traumatic Stress Disorder (in remission), and Substance Use Disorder (in remission, mild subtype).
* DSM-5 diagnoses of Cluster B Personality disorders.
* Positive urine drug screen for cocaine, opioids, amphetamine, and benzodiazepines at any visit

Stimulant Use Disorder, Cocaine Subtype Subjects:

* DSM-5 diagnoses other than: Stimulant Use Disorder, Cannabis Use Disorder, Alcohol Use Disorder (Mild Subtype), and Tobacco Use Disorder, Substance Induced Mood Disorder, Major Depressive Disorder (in remission), Generalized Anxiety Disorder (in remission), Post-Traumatic Stress Disorder (in remission).
* DSM-5 diagnoses of Cluster B Personality Disorders.
* Positive urine drug screen for opioids, amphetamine, and benzodiazepines at any visit

ADHD Subjects:

* DSM-5 diagnoses other than ADHD, Substance Induced Mood Disorder, Major Depressive Disorder (in remission), Generalized Anxiety Disorder (in remission), Post-Traumatic Stress Disorder (in remission), Substance Use Disorder (mild subtype, in remission).
* DSM-5 diagnoses of Cluster B Personality Disorders.
* Stimulant medication taken the morning of behavioral testing.
* Positive urine drug screen for cannabis, cocaine, opioids, amphetamine, methamphetamine or benzodiazepines at any visit. Subjects with a valid prescription for amphetamines for the treatment of ADHD will not be excluded.
* Unable or unwilling to withhold medications prescribed for treatment of ADHD on the morning of any behavioral testing clinic visit.
* Further exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: subjects meeting criteria for one of the described cohorts
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2016-07-22 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2018-09-06 (Actual)

PRIMARY OUTCOMES:
Stability in scores measured as change from baseline to follow-up visit at 4 (+/-1) weeks for Go/No Go Task | up to 5 weeks
Stability in scores measured as change from baseline to follow-up visit at 4 (+/-1) weeks for Stop Signal Reaction Time (SSRT) Task | up to 5 weeks
Stability in scores measured as change from baseline to follow-up visit at 4 (+/-1) weeks for Computerized Monetary Choice Task | up to 5 weeks
Stability in scores measured as change from baseline to follow-up visit at 4 (+/-1) weeks for Barratt Impulsiveness Questionnaire version 11 (BIS-11) | up to 5 weeks
Stability in scores measured as change from baseline to follow-up visit at 4 (+/-1) weeks for Immediate Memory Task (IMT) | up to 5 weeks
Stability in scores measured as change from baseline to follow-up visit at 4 (+/-1) weeks for Urgency, Premeditation, Perseverance, Sensation Seeking and Positive Urgency (UPPs-P) Impulsive Behavior Scale | up to 5 weeks

SECONDARY OUTCOMES:
Antisaccade performance measured as change from baseline to follow-up visit at 4 (+/-1) weeks on the eye tracker | up to 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States